CLINICAL TRIAL: NCT01693640
Title: A Pilot Study of the Safety and Efficacy of Abatacept Injections in the Treatment of Mucocutaneous Manifestations of Behcet's Syndrome
Brief Title: A Pilot Study of the Safety and Efficacy of Abatacept Injections in the Treatment of Behcet's Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-02611
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Female Patients With Behcet's Syndrome
Keywords: Behcet's
MeSH Terms: conditions — Behcet Syndrome | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- abatacept (Experimental)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Weekly injections with Abatacept 125 mg over 6 months
  Other Names: Orencia

SUMMARY:
Hypothesis: Abatacept injections will decrease the number of oral ulcers seen in Behcet's patients

DETAILED DESCRIPTION:
This will be an open label study, where 20 Behcet's patients with resistant oral ulcers and 10 with resistant genital ulcers will be enrolled (screen 40). After enrollment all patients will be followed for a month to document the number of oral and genital ulcers on their current regimen. Then all patients will receive abatacept for 6 months (evaluated at weeks 0, 2, 4, 8, 12, 16 and 24). Then the treatment will be stopped and they will be observed for the next 2 months, for a total of 9 month trial.

ELIGIBILITY:
Inclusion Criteria

1. Before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel.
2. Female patients with a diagnosis of Behcet's syndrome
3. Women, greater than 18 years of age
4. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 10 weeks after the last dose of study drug to minimize the risk of pregnancy.
5. Patients must have oral ulcers or genital ulcers that have been resistant to colchicine or topical measures for at least a month.

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 10 weeks after the last dose of study drug.
2. Women who are pregnant or breastfeeding.
3. Women with a positive pregnancy test on enrollment or before administration of abatacept.

   Target Disease Exceptions [Include as applicable]
   * Any patients with systemic manifestations of Behcet's syndrome (Patients with eye, CNS, vascular involvement, gastrointestinal disease)
   * Patients who are already on other immunosuppressive medications (azathioprine, TNF inhibitors, other biologic agents, methotrexate, mycophenolate mofetil, cyclosporine, cyclophosphamide)
4. Subjects who are impaired, incapacitated, or incapable of completing study-related assessments.
5. Subjects with current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic, or cerebral disease, whether or not related to Behcet's syndrome and which, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
6. Female subjects who have had a breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory, or other diagnostic evaluations.
7. Subjects with a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ.
8. Subjects who currently abuse drugs or alcohol.
9. Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of human immunodeficiency virus (HIV) detected during screening.
10. Subjects with herpes zoster or cytomegalovirus (CMV) that resolved less than 2 months before the informed consent document was signed.
11. Subjects who have received any live vaccines within 3 months of the anticipated first dose of study medication.
12. Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any chronic bacterial infection (eg, chronic pyelonephritis, osteomyelitis, or bronchiectasis).
13. Subjects at risk for tuberculosis (TB).
14. Subjects must not be positive for hepatitis B surface antigen.
15. Subjects who are positive for hepatitis C antibody if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay.
16. Subjects with any of the following laboratory values
17. Hemoglobin < 8.5 g/dL
18. WBC < 3000/mm3 (< 3 x 109/L)
19. Platelets < 100,000/mm3 (< 3 x 109/L)
20. Serum creatinine > 2 times the ULN
21. Serum ALT or AST > 2 times the ULN
22. Any other laboratory test results that, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
23. Subjects who have at any time received treatment with any investigational drug within 28 days (or less than 5 terminal half-lives of elimination) of the Day 1 dose.
24. Any concomitant biologic DMARD.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
ulcers | 6 month treatment period
  The primary endpoint is number of oral and genital ulcers (AUC) during the treatment period

SECONDARY OUTCOMES:
Genital ulcers | 6 month treatment
  Number of genital ulcers
Treatment failures | 6 months
  Number of patients who fail to complete 6 months (treatment failures)
Oral ulcer pain | 6 months
  Oral ulcer pain-Visual Analog Scale (VAS)
Side Effects | 6 months
  Monitoring of side effects
MDHAQ | 6 months
  Multidimensional health assessment questionnaire (MDHAQ)
BSAS | 6 months
  Behcet's syndrome activity score (BSAS)
BDCAF | 6 months
  Behcet's disease current activity form (BDCAF) scores

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Center for Musculoskeletal Care, New York, New York, United States

REFERENCES:
- See also: NYU Center for Musculoskeletal Care — http://redaf.med.nyu.edu/musculoskeletal-institute-%E2%80%93-333-east-38th-street